CLINICAL TRIAL: NCT05409430
Title: Prospective, Single-arm, Multi-center Study to Confirm the Safety and Performance of the ANA 5F Advanced Neurovascular Access®, in Combination With a Stent Retriever in Patients With Acute Ischemic Stroke (ANAIS)
Brief Title: ANAIS Study to Confirm the Safety and Performance of the ANA 5F Advanced Neurovascular Access®
Acronym: ANAIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anaconda Biomed S.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANA2201
Record Dates: First submitted 2022-05-31; First posted 2022-06-08 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Acute Ischemic Stroke
Keywords: AIS
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: Patients with Acute Ischemic Stroke (AIS), indicated for treatment with ANA 5F device in combination with Solitaire stent retriever, whose stroke is attributable to an occlusion of a large artery in the neurovasculature.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with Acute Ischemic Stroke (AIS) (Experimental): Patients with Acute Ischemic Stroke (AIS), indicated for treatment with ANA 5F device in combination with Solitaire stent retriever, whose stroke is attributable to an occlusion of a large artery in the neurovasculature.
  Interventions: Device: Neurothrombectomy

INTERVENTIONS:
Device: Neurothrombectomy — The ANA 5F device is intended to be inserted, be navigated to the neurovascular anatomy inside an outer catheter and be used as a conduit for insertion and guidance of intravascular catheters and retrieval devices into a selected blood vessel. The funnel is deployed by retracting the conduit catheter and is intended, when deployed, to provide temporary vascular flow restriction.
  The device is indicated for the introduction of interventional devices into the neuro vasculature, during interventions for restoring blood flow in patients experiencing acute ischemic stroke due to large vessel occlusion.
  Other Names: Mechanical thrombectomy (MT)

SUMMARY:
Prospective, single-arm, multi-center study to assess the safety and performance of the ANA 5F Advanced Neurovascular Access®, in combination with a stent retriever in patients with acute ischemic stroke.

DETAILED DESCRIPTION:
ANA 5F Advanced Neurovascular Access®: distal access catheter system designed to assist in neurovascular procedures by facilitating the insertion and guidance of other devices (i.e. retrieval devices and intravascular catheters) and temporarily restricting blood flow at the target position.

The objective of this study is to confirm the safety and performance of the ANA 5F device to be used as a tool to facilitate the Solitaire stent retriever placement and provide temporary restriction of blood flow in stroke patients undergoing neurothrombectomy for an acute large vessel occlusion (LVO) treated 24 hours from symptom onset (last time the subject was seen well).

Population: Up to 30 Participants with Acute Ischemic Stroke (AIS), indicated for treatment with ANA 5F device in combination with Solitaire stent retriever, whose stroke is attributable to an occlusion of a large artery in the neurovasculature.

ELIGIBILITY:
Inclusion Criteria:

* Clinical

  1. Age ≥18 and ≤85 years.
  2. Informed consent obtained from subject or acceptable subject surrogate (i.e. next of kin, or legal representative).
  3. A new focal disabling neurologic deficit consistent with acute cerebral ischemia.
  4. Baseline NIHSS obtained prior to procedure ≥ 8 points and ≤ 25 points.
  5. Pre-ictal mRS score of 0 or 1.
  6. Treatable as soon as possible and at least within 24 hours of symptom onset, defined as point in time when the subject was last seen well (at baseline) (Treatment start is defined as access puncture).
  7. Subjects being either (1) eligible for, and received, IV tPA/TNK within 3 hours of symptom onset or (2) ineligible for IV tPA/TNK treatment.

     Neuro Imaging
  8. Occlusion (TICI 0 or TICI 1 flow), of the terminal internal carotid artery, M1 or M2 segments of the middle cerebral artery, suitable for mechanical embolectomy, confirmed on conventional angiography.
  9. For patients treated ≤ 6 hours:

     1. MRI criterion: volume of diffusion restriction visually assessed ≤50 mL

        OR
     2. CT criterion: Alberta Stroke program early CT score (ASPECTS) 6 to 10 on baseline CT.

     For patients treated 6 to 24 hours. Target Mismatch Profile on CT perfusion or MRI (ischemic core volume is < 70 ml, mismatch ratio is > 1.8 and mismatch volume is > 15 ml)
  10. The subject is indicated for neurothrombectomy treatment with SOLITAIRE, by the Interventionalist.

Exclusion Criteria:

* Clinical

  1. Initially treated with a different thrombectomy device.
  2. Subject has suffered a stroke in the past 1 year.
  3. Occlusion (TICI 0 or TICI 1 flow) of the basilar or vertebral arteries.
  4. Clinical symptoms suggestive of bilateral stroke or stroke in multiple territories.
  5. Known hemorrhagic diathesis, coagulation factor deficiency, or oral anticoagulant therapy with antivitamin K, with INR >3.0.
  6. Known baseline glucose of <50 mg/dL or >400 mg/dL.
  7. Severe, sustained hypertension (systolic blood pressure >185 mmHg or diastolic blood pressure >110 mmHg).
  8. Serious, advanced, or terminal illness with anticipated life expectancy of less than 1 year.
  9. History of life-threatening allergy (more than rash) to contrast medium.
  10. Known renal insufficiency with creatinine ≥3 mg/dL or Glomerular Filtration Rate (GFR) <30 mL/min.
  11. Cerebral vasculitis.
  12. Subject is a current user or has a recent history of cocaine use.
  13. Pregnant and/or lactating woman.
  14. Patient participating in a study involving an investigational drug or device that would impact this study.
  15. Patients that are unlikely to be available for a 90-day follow-up (e.g. no fixed home address, visitor from overseas).

      Neuro Imaging
  16. CT or MRI evidence of hemorrhage (the presence of microbleeds is allowed).
  17. Angiographic evidence of vasculitis.
  18. Significant mass effect with midline shift.
  19. Evidence of complete occlusion, high grade stenosis or arterial dissection in the extracranial or internal carotid artery (ICA).
  20. Subjects with known or suspected underlying intracranial atherosclerotic lesions responsible for the target occlusion.
  21. Subjects with occlusions in multiple vascular territories (e.g., bilateral anterior circulation, or anterior/posterior circulation).
  22. Evidence of intracranial tumor.
  23. Suspicion of aortic dissection presumed septic embolus, or suspicion of bacterial endocarditis.
  24. Severe arterial tortuosity likely to prevent stable positioning of the guide catheter in the distal cervical segment (C1) or petrous segment (C2) of internal carotid artery (ICA).

      Technical
  25. Inability to create an arterial access and / or to advance a guide catheter due to anatomical or physiological restrictions (i.e. vasospasm).
  26. Inability of the guide catheter to obtain a stable position in the ICA.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2023-07-10 (Actual)

PRIMARY OUTCOMES:
Successful reperfusion, defined as rate of patients achieving mTICI ≥2b. | Day0. Intraoperative
  Successful reperfusion, defined as rate of patients achieving mTICI ≥2b in the target vessel within three passes of the ANA 5F before the use of rescue therapy, assessed by the Core Lab.
The composite of symptomatic Intracranial Hemorrhage (sICH) within 24 hours (-8 / +12 h) post-procedure, together with serious adverse device effects. | 24 hours (-8 / +12 h) post-procedure
  The composite of symptomatic Intracranial Hemorrhage (sICH) within 24 hours (-8 / +12 h) post-procedure, together with serious adverse device effects (excluding those already counted in sICH) at Day 5 (± 12 h) or discharge (whatever comes first).

SECONDARY OUTCOMES:
Occurrence of Intracranial Hemorrhage (ICH); any symptomatic or asymptomatic ICH | 90 days

OTHER OUTCOMES:
Rate of subjects with a neurological deterioration of ≥4 points on NIHSS | 24 hours
Occurrence of embolization in a previously uninvolved territory on the cerebral angiogram. | Day 0. Intraoperative
Procedure-related mortality rate. | Day 5 (± 12 hours) or discharge, whichever comes first, and at 90 days.

CONTACTS AND LOCATIONS:
Overall Officials: René Spaargaren, MD, Study Chair — Anaconda Biomed S.L.
Locations (3):
- Spain (3):
  - Hospital Universitari de la Vall d'Hebron, Barcelona
  - Hospital Universitari Dr. Josep Trueta, Girona
  - Hospital Clínico Universitario Virgen de la Arrixaca, Murcia

IPD SHARING:
Plan to Share IPD: Undecided